CLINICAL TRIAL: NCT04976192
Title: Study to Evaluate the Efficacy, Safety, Tolerability, and Immunogenicity of TEV-45779 Compared to XOLAIR (Omalizumab) in Patients With Chronic Idiopathic/Spontaneous Urticaria Who Remain Symptomatic Despite Antihistamine (H1) Treatment.
Brief Title: Study to Compare Efficacy and Safety of TEV-45779 With XOLAIR (Omalizumab) in Adults With Chronic Idiopathic Urticaria
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Teva Pharmaceuticals USA (Industry)
Collaborators: Teva Pharmaceuticals Development, Inc. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TV45779-IMB-30086; 2021-001796-17 (EudraCT Number)
Record Dates: First submitted 2021-07-14; First posted 2021-07-26 (Actual); Results first posted 2025-10-07 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-09

CONDITIONS: Chronic Urticaria
MeSH Terms: conditions — Chronic Urticaria | interventions — Omalizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (10):
- TEV-45779-300 mg Main Treatment period (Experimental): TEV-45779 (Omalizumab) injection 150 mg/mL pre-filled syringe administered twice (total dosage 300 mg) at week 0, 4, 8
  Interventions: Combination Product: TEV-45779
- Xolair-300 mg Main Treatment Period (Active Comparator): XOLAIR (omalizumab) injection 150 mg/mL pre-filled syringe administered twice (total dosage 300 mg) at week 0, 4, 8
  Interventions: Combination Product: XOLAIR® Injection
- TEV-45779-150 mg Main Treatment period (Experimental): TEV-45779 (Omalizumab) injection 150 mg/mL pre-filled syringe administered with one placebo injection at week 0, 4, 8
  Interventions: Combination Product: TEV-45779
- Xolair-150 mg Main Treatment Period (Active Comparator): XOLAIR (omalizumab) injection 150 mg/mL pre-filled syringe administered with one placebo injection at week 0, 4, 8
  Interventions: Combination Product: XOLAIR® Injection
- TEV-45779-300 mg Main / TEV45779-300 mg Transition Period (Experimental): TEV-45779 (Omalizumab) injection 150 mg/mL pre-filled syringe administered twice (total dosage 300 mg) at week 12,16,20 in patients that were randomized to TEV-45779-300 mg in the Main Treatment period.
  Interventions: Combination Product: TEV-45779
- Xolair-300 mg Main / TEV45779-300 mg Transition Period (Experimental): TEV-45779 (Omalizumab) injection 150 mg/mL pre-filled syringe administered twice (total dosage 300 mg) at week 12,16,20 in patients that were randomized to Xolair-300 mg in the main treatment period.
  Interventions: Combination Product: TEV-45779; Combination Product: XOLAIR® Injection
- Xolair-300 mg Main / Xolair-300 mg Transition Period (Active Comparator): XOLAIR (omalizumab) injection 150 mg/mL pre-filled syringe administered twice (total dosage 300 mg) at week 12,16,20 in patients that were randomized to Xolair-300 mg in the main treatment period.
  Interventions: Combination Product: XOLAIR® Injection
- TEV-45779-150 mg Main / TEV-45779-150 mg Transition Period (Experimental): TEV-45779 (Omalizumab) injection 150 mg/mL pre-filled syringe administered with one placebo injection at week 12,16,20 in patients that were randomized to TEV-45779-150 mg in the main treatment period.
  Interventions: Combination Product: TEV-45779
- Xolair-150 mg Main / TEV-45779-150 mg Transition Period (Experimental): TEV-45779 (Omalizumab) injection 150 mg/mL pre-filled syringe administered with one placebo injection at week 12,16,20 in patients that were randomized to XOLAIR-150 mg in the main treatment period.
  Interventions: Combination Product: TEV-45779; Combination Product: XOLAIR® Injection
- Xolair-150 mg Main / Xolair-150 mg Transition Period (Active Comparator): XOLAIR (omalizumab) injection 150 mg/mL pre-filled syringe administered with one placebo injection at week 12,16,20 in patients that were randomized to XOLAIR -150 mg in the main treatment period.
  Interventions: Combination Product: XOLAIR® Injection

INTERVENTIONS:
Combination Product: TEV-45779 — TEV-45779 (Omalizumab) solution for injection 150 mg/mL prefilled syringe
  Arms: TEV-45779-150 mg Main / TEV-45779-150 mg Transition Period; TEV-45779-150 mg Main Treatment period; TEV-45779-300 mg Main / TEV45779-300 mg Transition Period; TEV-45779-300 mg Main Treatment period; Xolair-150 mg Main / TEV-45779-150 mg Transition Period; Xolair-300 mg Main / TEV45779-300 mg Transition Period
Combination Product: XOLAIR® Injection — XOLAIR (omalizumab) injection is supplied as a single dose PFS. Each PFS of XOLAIR contains 150 mg of omalizumab in 1 mL of solution.
  Arms: Xolair-150 mg Main / TEV-45779-150 mg Transition Period; Xolair-150 mg Main / Xolair-150 mg Transition Period; Xolair-150 mg Main Treatment Period; Xolair-300 mg Main / TEV45779-300 mg Transition Period; Xolair-300 mg Main / Xolair-300 mg Transition Period; Xolair-300 mg Main Treatment Period

SUMMARY:
The purpose of the study is to compare the efficacy, pharmacokinetics, pharmacodynamics, safety, tolerability, and immunogenicity of TEV-45779 compared to XOLAIR in patients with Urticaria (CIU)/Chronic Spontaneous Urticaria (CSU) who remain symptomatic on H1 antihistamine treatment.

DETAILED DESCRIPTION:
This is a multicenter, randomized, double-blind study to demonstrate similar efficacy and safety of TEV-45779 compared to XOLAIR administered sc at doses of 300 mg or 150 mg every 4 weeks for 24 weeks (6 treatments) in patients with Chronic Idiopathic Urticaria (CIU)/Chronic Spontaneous Urticaria (CSU) who remain symptomatic despite antihistamine (H1) treatment. This study will consist of a screening period (up to 2 weeks), a 24-week treatment period consisting of a 12-week double-blind main treatment period and a 12-week double-blind transition period, which is followed by a 16-week follow-up period. The total duration of the study is up to 42 weeks.

At baseline, patients will be randomized in a 2:2:1:1 ratio to receive the first 3 treatments of TEV-45779 300 mg, XOLAIR 300 mg, TEV-45779 150 mg or XOLAIR 150 mg (main treatment period). At Week 12, prior to receiving their fourth dose of study medication, patients in the XOLAIR 300 mg and the XOLAIR 150 mg treatment groups will be randomized 1:1 to receive 3 additional doses of XOLAIR (at the same dose level as prior to randomization, or switch to 3 doses of TEV-45779 (transition period) at the same dose level as prior to randomization. All patients in the TEV-45779 groups will continue to receive TEV-45779 at the same dose levels.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of CIU refractory to H1 antihistamines for ≥3 months

Exclusion Criteria:

* Chronic urticaria with clearly defined underlying etiology
* Other skin disease associated with itch
* Evidence of parasitic infection on stool evaluation for ova and parasites
* History of anaphylactic shock
* Hypersensitivity to omalizumab or any component of the formulation
* Required background therapy with other than protocol-defined antihistamines
* Any medical condition that could jeopardize or would compromise the patient's safety or ability to participate in this study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 608 (Actual)
Dates: Start 2021-08-30 (Actual); Primary Completion 2024-04-05 (Actual); Study Completion 2024-04-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Teva Medical Expert, MD, Study Director — Teva Pharmaceuticals Development, Inc.
Locations (9):
- United States (9):
  - 10008, Bakersfield, California
  - Site 10001, Clearwater, Florida
  - 10012, Coral Gables, Florida
  - 10006, Kissimmee, Florida
  - 10014, Maitland, Florida
  - 10005, Miami, Florida
  - 10009, Tampa, Florida
  - 10007, Troy, Michigan
  - 10004, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study included a 24-week treatment period consisting of a 12-week double-blind main treatment period and a 12-week double-blind transition period, which was followed by a 16-week follow-up period.
Groups:
- Main Treatment Period: TEV-45779 High Dose: Participants received TEV-45779 subcutaneous (SC) injection at a high dose level every 4 weeks (Q4W) at Weeks 0, 4, and 8.
- Main Treatment Period: TEV-45779 Low Dose: Participants received TEV-45779 SC injection at a low dose level Q4W at Weeks 0, 4, and 8.
- Main Treatment Period: XOLAIR High Dose: Participants received XOLAIR SC injection at a high dose level Q4W at Weeks 0, 4, and 8.
- Main Treatment Period: XOLAIR Low Dose: Participants received XOLAIR SC injection at a low dose level Q4W at Weeks 0, 4, and 8.
- Transition Period: TEV-45779/TEV-45779 High Dose: Participants who received TEV-45779 SC injection at a high dose level in the main treatment period, continued to receive TEV-45779 at the same dose level at Weeks 12, 16, and 20 in the transition period.
- Transition Period: TEV-45779/TEV-45779 Low Dose: Participants who received TEV-45779 SC injection at a low dose level in the main treatment period, continued to receive TEV-45779 at the same dose level at Weeks 12, 16, and 20 in the transition period.
- Transition Period: XOLAIR/XOLAIR High Dose: Participants who received XOLAIR SC injection at a high dose level in the main treatment period, continued to receive XOLAIR at the same dose level at Weeks 12, 16, and 20 in the transition period.
- Transition Period: XOLAIR/XOLAIR Low Dose: Participants who received XOLAIR SC injection at a low dose level in the main treatment period, continued to receive XOLAIR at the same dose level at Weeks 12, 16, and 20 in the transition period.
- Transition Period: XOLAIR/TEV-45779 High Dose: Participants who received XOLAIR SC injection at a high dose level in the main treatment period, received TEV-45779 SC injection at a high dose level at Weeks 12, 16, and 20 in the transition period.
- Transition Period: XOLAIR/TEV-45779 Low Dose: Participants who received XOLAIR SC injection at a low dose level in the main treatment period, received TEV-45779 SC injection at a low dose level at Weeks 12, 16, and 20 in the transition period.
Period: Main Treatment Period (12 Weeks)
Arm/Group | Main Treatment Period: TEV-45779 High Dose | Main Treatment Period: TEV-45779 Low Dose | Main Treatment Period: XOLAIR High Dose | Main Treatment Period: XOLAIR Low Dose | Transition Period: TEV-45779/TEV-45779 High Dose | Transition Period: TEV-45779/TEV-45779 Low Dose | Transition Period: XOLAIR/XOLAIR High Dose | Transition Period: XOLAIR/XOLAIR Low Dose | Transition Period: XOLAIR/TEV-45779 High Dose | Transition Period: XOLAIR/TEV-45779 Low Dose
Started | 201 | 102 | 203 | 102 | 0 | 0 | 0 | 0 | 0 | 0
Received at Least 1 Dose of Study Drug | 201 | 102 | 203 | 102 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 188 | 98 | 194 | 101 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 13 | 4 | 9 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 12 | 3 | 8 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Other Than Specified | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Transition Treatment Period (12 Weeks)
Arm/Group | Main Treatment Period: TEV-45779 High Dose | Main Treatment Period: TEV-45779 Low Dose | Main Treatment Period: XOLAIR High Dose | Main Treatment Period: XOLAIR Low Dose | Transition Period: TEV-45779/TEV-45779 High Dose | Transition Period: TEV-45779/TEV-45779 Low Dose | Transition Period: XOLAIR/XOLAIR High Dose | Transition Period: XOLAIR/XOLAIR Low Dose | Transition Period: XOLAIR/TEV-45779 High Dose | Transition Period: XOLAIR/TEV-45779 Low Dose
Started | 0 | 0 | 0 | 0 | 188 | 98 | 97 | 51 | 97 | 50
Received at Least 1 Dose of Study Drug | 0 | 0 | 0 | 0 | 188 | 98 | 97 | 51 | 97 | 50
Completed | 0 | 0 | 0 | 0 | 178 | 90 | 93 | 49 | 95 | 47
Not Completed | 0 | 0 | 0 | 0 | 10 | 8 | 4 | 2 | 2 | 3
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 9 | 7 | 4 | 2 | 2 | 3
Not completed — Other Than Specified | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The intent-to-treat (ITT) analysis set included all randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Main Treatment Period: TEV-45779 High Dose | Main Treatment Period: TEV-45779 Low Dose | Main Treatment Period: XOLAIR High Dose | Main Treatment Period: XOLAIR Low Dose | Total
Number analyzed (Participants) | 201 | 102 | 203 | 102 | 608
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.1 (14.30) | 42.7 (13.64) | 42.0 (13.75) | 41.5 (14.29) | 41.7 (13.99)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 132 | 69 | 138 | 67 | 406
  Male | 69 | 33 | 65 | 35 | 202
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 45 | 13 | 26 | 11 | 95
  Not Hispanic or Latino | 153 | 88 | 174 | 89 | 504
  Unknown or Not Reported | 3 | 1 | 3 | 2 | 9
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: American Indian/Alaskan/Native American | 12 | 4 | 4 | 0 | 20
  Race: Asian | 65 | 35 | 75 | 38 | 213
  Race: Black/African American | 0 | 3 | 2 | 0 | 5
  Race: White | 123 | 59 | 118 | 61 | 361
  Race: Other/Mixed | 1 | 0 | 3 | 2 | 6
  Race: Not Reported/Unknown | 0 | 1 | 1 | 1 | 3
Weekly Itch Severity Score (ISS7) [Mean (Standard Deviation); unit: units on a scale] — Severity of itch was recorded by participants twice daily in their eDiary, on a scale of 0 (none) to 3 (intense/severe). A weekly score (ISS7) was defined as the sum of available daily itch severity scores in that week, divided by the number of days for which a daily itch severity score was available, multiplied by 7. The daily ISS was was calculated as the average of the morning and evening scores. The possible range of weekly score was therefore 0 (best score) to 21 (worst score) with higher scores indicating more severe itching. Population: Here, 'number analyzed' = participants evaluable at Baseline for this baseline characteristic.
  units on a scale
    number analyzed (Participants) | 196 | 100 | 203 | 102 | 601
    (all) | 16.26 (3.721) | 16.14 (3.361) | 16.28 (3.524) | 16.00 (3.723) | 16.20 (3.590)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the ISS7 at Week 12, TEV-45779 High Dose Compared to XOLAIR High Dose (For European Medicines Agency [EMA] Submission)
Description: The severity of the itch was recorded by the participants twice daily in their eDiary, on a scale of 0 (none) to 3 (intense/severe). A weekly itch score (ISS7) was defined as the sum of the available daily itch severity scores in that week, divided by the number of days for which a daily itch severity score was available, multiplied by 7. The daily ISS was calculated as the average of the morning and evening scores. The possible range of the weekly score was therefore 0 (best score) to 21 (worst score) with higher scores indicating more severe itching. Least square (LS) mean and 95% confidence interval (CI) were calculated using analysis of covariance (ANCOVA) model. Multiple imputation performed both for the participants having missing ISS7 at week 12 and for participants using any disallowed concomitant medication.
Time Frame: Baseline, Week 12
Population: The ITT analysis set included all randomized participants.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Main Treatment Period: TEV-45779 High Dose | Main Treatment Period: XOLAIR High Dose
Number analyzed (Participants) | 201 | 203
units on a scale | -10.92 (-11.85) [-11.85 to -9.99] | -10.61 (-11.51) [-11.51 to -9.71]
Statistical Analysis 1: Comparison: Main Treatment Period: TEV-45779 High Dose vs Main Treatment Period: XOLAIR High Dose; Test type: Other; LS Mean Difference = -0.31, 95% CI 2-sided [-1.56 to 0.94]

2. Primary Outcome: Change From Baseline in the ISS7 at Week 12, TEV-45779 High Dose Compared to XOLAIR High Dose (For Food and Drug Administration [FDA] Submission)
Description: The severity of the itch was recorded by the participants twice daily in their eDiary, on a scale of 0 (none) to 3 (intense/severe). A weekly itch score (ISS7) was defined as the sum of the available daily itch severity scores in that week, divided by the number of days for which a daily itch severity score was available, multiplied by 7. The daily ISS was calculated as the average of the morning and evening scores. The possible range of the weekly score was therefore 0 (best score) to 21 (worst score) with higher scores indicating more severe itching. LS mean and 90% CI were calculated using ANCOVA model. Multiple imputation performed for the participants having missing ISS7 at week 12.
Time Frame: Baseline, Week 12
Population: The ITT analysis set included all randomized participants.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Main Treatment Period: TEV-45779 High Dose | Main Treatment Period: XOLAIR High Dose
Number analyzed (Participants) | 201 | 203
units on a scale | -10.77 [-11.61 to -9.93] | -10.38 [-11.24 to -9.52]
Statistical Analysis 1: Comparison: Main Treatment Period: TEV-45779 High Dose vs Main Treatment Period: XOLAIR High Dose; Test type: Other; LS Mean Difference = -0.39, 90% CI 2-sided [-1.37 to 0.58]
Statistical Analysis 2: Comparison: Main Treatment Period: TEV-45779 High Dose vs Main Treatment Period: XOLAIR High Dose; The relative potency of the test drug to the reference drug was defined as the dose of the test drug that produced the same biological response as 1 unit of the dose of the reference drug. Relative potency was demonstrated if the 90% confidence interval (CI) for relative potency fell entirely within the equivalence margins; Test type: Other; Relative Potency = 0.89 — Relative potency of TEV-45779 and XOLAIR is a co-primary efficacy endpoint for FDA submission

3. Secondary Outcome: Change From Baseline in the ISS7 at Weeks 4 and 12
Description: The severity of the itch was recorded by the participants twice daily in their eDiary, on a scale of 0 (none) to 3 (intense/severe). A weekly itch score (ISS7) was defined as the sum of the available daily itch severity scores in that week, divided by the number of days for which a daily itch severity score was available, multiplied by 7. The daily ISS was calculated as the average of the morning and evening scores. The possible range of the weekly score was therefore 0 (best score) to 21 (worst score) with higher scores indicating more severe itching. The observed mean and standard deviation values are reported here with no imputation performed.
Time Frame: Baseline, Weeks 4 and 12
Population: The ITT analysis set included all randomized participants. 'Overall number of participants analyzed' = participants evaluable for this endpoint. 'Number analyzed' = participants evaluable at specified timepoint.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Main Treatment Period: TEV-45779 High Dose | Main Treatment Period: TEV-45779 Low Dose | Main Treatment Period: XOLAIR High Dose | Main Treatment Period: XOLAIR Low Dose
Number analyzed (Participants) | 192 | 98 | 198 | 97
units on a scale
  Change at Week 4 | -7.64 (6.383) | -7.35 (6.236) | -7.87 (6.033) | -7.27 (6.084)
  Change at Week 12: number analyzed (Participants) | 184 | 96 | 196 | 97
  Change at Week 12 | -10.92 (6.512) | -9.96 (6.340) | -10.65 (6.490) | -10.35 (6.082)

4. Secondary Outcome: Change From Baseline in Weekly Urticaria Activity Score (UAS7) at Week 12
Description: The UAS was a composite eDiary-recorded score with numeric severity intensity ratings on a scale of 0 - 3 (0 = none to 3 = intense/severe) for (1) the number of wheals (hives); and (2) the intensity of the itch separately, measured twice daily (morning and evening). The daily UAS was the average of the morning and evening scores, which ranged from 0 (none) to 6 (severe). The UAS7 was the sum of the daily UAS scores over 7 days, which ranged from 0 (minimum) to 42 (highest urticaria severity). Higher scores indicated greater severity of urticaria symptoms.
Time Frame: Baseline, Week 12
Population: The ITT analysis set included all randomized participants. 'Overall number of participants analyzed' = participants evaluable for this endpoint.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Main Treatment Period: TEV-45779 High Dose | Main Treatment Period: TEV-45779 Low Dose | Main Treatment Period: XOLAIR High Dose | Main Treatment Period: XOLAIR Low Dose
Number analyzed (Participants) | 184 | 96 | 196 | 97
units on a scale | -22.10 (13.204) [lower limit 13.204] | -20.67 (12.223) [lower limit 12.223] | -21.73 (12.651) [lower limit 12.651] | -21.67 (12.158) [lower limit 12.158]

5. Secondary Outcome: Percentage of Participants With a UAS7 Score ≤6 at Week 12
Description: The UAS was a composite eDiary-recorded score with numeric severity intensity ratings on a scale of 0 - 3 (0 = none to 3 = intense/severe) for (1) the number of wheals (hives); and (2) the intensity of the itch separately, measured twice daily (morning and evening). The daily UAS was the average of the morning and evening scores, which ranged from 0 (none) to 6 (severe). The UAS7 is the number of participants achieving the endpoint of less than or equal to 6. UAS7 was calculated as the sum of the daily UAS scores over 7 days, which ranged from 0 (minimum) to 42 (highest urticaria severity). Higher scores indicated greater severity of urticaria symptoms.
Time Frame: Week 12
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Main Treatment Period: TEV-45779 High Dose | Main Treatment Period: TEV-45779 Low Dose | Main Treatment Period: XOLAIR High Dose | Main Treatment Period: XOLAIR Low Dose
Number analyzed (Participants) | 184 | 96 | 196 | 97
percentage of participants | 49.5 | 45.8 | 46.4 | 48.5

6. Secondary Outcome: Percentage of Complete Responders (UAS7 Score = 0) at Week 12
Description: The UAS was a composite eDiary-recorded score with numeric severity intensity ratings on a scale of 0 - 3 (0 = none to 3 = intense/severe) for (1) the number of wheals (hives); and (2) the intensity of the itch separately, measured twice daily (morning and evening). The daily UAS was the average of the morning and evening scores, which ranged from 0 (none) to 6 (severe). The UAS7 was the sum of the daily UAS scores over 7 days, which ranged from 0 (minimum) to 42 (highest urticaria severity). Higher scores indicated greater severity of urticaria symptoms. Complete responders were participants with a UAS7 score = 0.
Time Frame: Week 12
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Main Treatment Period: TEV-45779 High Dose | Main Treatment Period: TEV-45779 Low Dose | Main Treatment Period: XOLAIR High Dose | Main Treatment Period: XOLAIR Low Dose
Number analyzed (Participants) | 184 | 96 | 196 | 97
percentage of participants | 33.2 | 28.1 | 29.6 | 30.9

7. Secondary Outcome: Change From Baseline in the Physician's (In-clinic) Assessment of UAS at Week 12
Description: Physician's (in-clinic) assessment of UAS score was performed using the in-clinic UAS. The physician, or the person designated, provided the sum of the score of the participant's urticaria lesions (number of wheals [hives]) and pruritus (itch) reflective of the participant's condition over the 12 hours prior to the visit using the rating scale of 0 - 6 (0 = none to 6 = intense/severe). Higher scores indicated greater severity of urticaria symptoms.
Time Frame: Baseline, Week 12
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Main Treatment Period: TEV-45779 High Dose | Main Treatment Period: TEV-45779 Low Dose | Main Treatment Period: XOLAIR High Dose | Main Treatment Period: XOLAIR Low Dose
Number analyzed (Participants) | 185 | 96 | 193 | 101
units on a scale | -3.38 (2.002) [lower limit 2.002] | -3.34 (1.907) [lower limit 1.907] | -3.55 (1.893) [lower limit 1.893] | -3.15 (2.085) [lower limit 2.085]

8. Secondary Outcome: Change From Baseline in the Weekly Number of Wheals Score at Week 12
Description: The wheals (hives) severity score, defined by number of wheals (hives), was recorded by the participant twice daily in their eDiary, on a scale of 0 (none) to 3 (> 12 hives/12 hours). A weekly number of wheals score was derived by adding up the average daily scores of the 7 days preceding the visit. The possible range of the weekly score was therefore 0 (no wheals) - 21 (highest hives activity).
Time Frame: Baseline, Week 12
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Main Treatment Period: TEV-45779 High Dose | Main Treatment Period: TEV-45779 Low Dose | Main Treatment Period: XOLAIR High Dose | Main Treatment Period: XOLAIR Low Dose
Number analyzed (Participants) | 184 | 96 | 196 | 97
units on a scale | -11.18 (7.127) [lower limit 7.127] | -10.70 (6.551) [lower limit 6.551] | -11.09 (6.740) [lower limit 6.740] | -11.33 (6.672) [lower limit 6.672]

9. Secondary Outcome: Change From Baseline in the Weekly Size of the Largest Wheals Score at Week 12
Description: The weekly size of the largest wheals score was calculated from the eDiary data. A wheal score of 0 was assigned when <10 small wheals (diameter <3 centimeters [cm]) were present, presence of 10-50 small wheals or less than 10 large wheals (diameter >3 cm) was denoted by score of 1. A score of 2 was assigned when more than 50 small wheals or 10 to 50 large wheals were present. A score of 3 denoted wheals covering almost the entire body surface area. A weekly score was defined as the sum of the available daily size of the largest wheals scores in that week, divided by the number of days for which a daily score was available, multiplied by 7. The possible range of the weekly score was therefore 0 (best score) to 21 (worst score) with higher scores indicating more severity.
Time Frame: Baseline, Week 12
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Main Treatment Period: TEV-45779 High Dose | Main Treatment Period: TEV-45779 Low Dose | Main Treatment Period: XOLAIR High Dose | Main Treatment Period: XOLAIR Low Dose
Number analyzed (Participants) | 184 | 96 | 196 | 97
units on a scale | -10.28 (6.937) [lower limit 6.937] | -9.52 (6.670) [lower limit 6.670] | -10.45 (6.745) [lower limit 6.745] | -10.68 (6.838) [lower limit 6.838]

10. Secondary Outcome: Time to Minimally Important Difference (MID) Response in ISS7 Score
Description: Time to MID response was defined as time to a reduction from baseline in ISS7 of ≥5 points in ISS7 score by Week 12.
Time Frame: Baseline up to Week 12
Population: The ITT analysis set included all randomized participants. 'Overall number of participants analyzed' = participants achieving MID up to Week 12.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Main Treatment Period: TEV-45779 High Dose | Main Treatment Period: TEV-45779 Low Dose | Main Treatment Period: XOLAIR High Dose | Main Treatment Period: XOLAIR Low Dose
Number analyzed (Participants) | 177 | 87 | 185 | 87
weeks | 2.0 [2.0 to 3.0] | 2.0 [1.0 to 2.0] | 2.0 [NA to NA] — Confidence interval for median time to MID could not be calculated (NA) because MID was reached too early in the observation period, resulting in an insufficient number of observations to calculate upper and lower limits. | 2.0 [2.0 to 3.0]

11. Secondary Outcome: Percentage of ISS7 MID Responders at Week 12
Description: A responder was defined as a participant with a reduction from baseline in ISS7 of ≥5 points in ISS7 score.
Time Frame: Week 12
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Main Treatment Period: TEV-45779 High Dose | Main Treatment Period: TEV-45779 Low Dose | Main Treatment Period: XOLAIR High Dose | Main Treatment Period: XOLAIR Low Dose
Number analyzed (Participants) | 184 | 96 | 196 | 97
percentage of participants | 81.0 | 78.1 | 80.6 | 79.4

12. Secondary Outcome: Percentage of Angioedema-Free Days From Week 4 to Week 12
Description: Percentage of angioedema-free days from Week 4 to Week 12 were calculated based on the diary data as the number of days in the diary between the dates of Week 4 and Week 12 visits with no angioedema episodes, divided by the total number of days with diary entries in this time span * 100%.
Time Frame: Week 4 to Week 12
Population: as for outcome 4
Measure: Median (Full Range); unit: percentage of days
Arm/Group | Main Treatment Period: TEV-45779 High Dose | Main Treatment Period: TEV-45779 Low Dose | Main Treatment Period: XOLAIR High Dose | Main Treatment Period: XOLAIR Low Dose
Number analyzed (Participants) | 195 | 99 | 202 | 102
percentage of days | 100.00 (0.0) [0.0 to 100.0] | 100.00 (0.0) [0.0 to 100.0] | 100.00 (0.0) [0.0 to 100.0] | 100.00 (0.0) [0.0 to 100.0]

13. Secondary Outcome: Change From Baseline in the Overall Dermatology Life Quality Index (DLQI) Score at Week 12
Description: The DLQI consisted of 10 questions concerning participants' perception of the impact of skin diseases on different aspects of their health-related quality of life over the last week. The DLQI total score was calculated by adding the score of each question (scored as follows: Very much = 3; Yes [in question 7.a] = 3; A lot = 2; A little = 1; Not at all = 0; Not relevant = 0; No [in question 7.a] = 0; Question unanswered = 0), resulting in a maximum of 30 and a minimum of 0. The higher the score, the more the quality of life was impaired. A score higher than 10 indicated that the participant's life was being severely affected by their skin disease.
Time Frame: Baseline, Week 12
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Main Treatment Period: TEV-45779 High Dose | Main Treatment Period: TEV-45779 Low Dose | Main Treatment Period: XOLAIR High Dose | Main Treatment Period: XOLAIR Low Dose
Number analyzed (Participants) | 188 | 98 | 193 | 100
units on a scale | -9.72 (7.125) [lower limit 7.125] | -8.40 (7.28) [lower limit 7.28] | -9.54 (7.091) [lower limit 7.091] | -8.09 (6.432) [lower limit 6.432]

14. Secondary Outcome: Change From Week 12 in ISS7 at Weeks 24 and 40
Description: The severity of the itch was recorded by the participants twice daily in their eDiary, on a scale of 0 (none) to 3 (intense/severe). A weekly itch score (ISS7) was defined as the sum of the available daily itch severity scores in that week, divided by the number of days for which a daily itch severity score was available, multiplied by 7. The daily ISS was calculated as the average of the morning and evening scores. The possible range of the weekly score was therefore 0 (best score) to 21 (worst score) with higher scores indicating more severe itching.
Time Frame: Week 12, Weeks 24 and 40
Population: The transition intent-to-treat (TITT) analysis set included all participants re-randomized in the transition period. 'Overall number of participants analyzed' = participants evaluable for this endpoint. 'Number analyzed' = participants evaluable at specified timepoint.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Transition Period: TEV-45779/TEV-45779 High Dose | Transition Period: TEV-45779/TEV-45779 Low Dose | Transition Period: XOLAIR/XOLAIR High Dose | Transition Period: XOLAIR/XOLAIR Low Dose | Transition Period: XOLAIR/TEV-45779 High Dose | Transition Period: XOLAIR/TEV-45779 Low Dose
Number analyzed (Participants) | 170 | 91 | 91 | 46 | 93 | 47
units on a scale
  Change at Week 24 | -1.64 (3.598) | -1.37 (4.576) | -1.82 (4.016) | -1.21 (3.186) | -1.78 (4.226) | -2.09 (4.585)
  Change at Week 40: number analyzed (Participants) | 145 | 75 | 75 | 39 | 83 | 39
  Change at Week 40 | 1.84 (7.182) | 0.44 (6.982) | 1.43 (6.870) | 1.58 (5.274) | 2.03 (7.969) | 1.27 (6.718)

15. Secondary Outcome: Change From Week 12 in the UAS7 at Week 24
Description: The UAS was a composite eDiary-recorded score with numeric severity intensity ratings on a scale of 0 - 3 (0 = none to 3 = intense/severe) for (1) the number of wheals (hives); and (2) the intensity of the itch separately, measured twice daily (morning and evening). The daily UAS was the average of the morning and evening scores, which can range from 0 (none) to 6 (severe). The UAS7 was the sum of the daily UAS scores over 7 days, which can range from 0 (minimum) to 42 (highest urticaria severity). Higher scores indicated greater severity of urticaria symptoms.
Time Frame: Week 12, Week 24
Population: The TITT analysis set included all participants re-randomized in the transition period. 'Overall number of participants analyzed' = participants evaluable for this endpoint.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Transition Period: TEV-45779/TEV-45779 High Dose | Transition Period: TEV-45779/TEV-45779 Low Dose | Transition Period: XOLAIR/XOLAIR High Dose | Transition Period: XOLAIR/XOLAIR Low Dose | Transition Period: XOLAIR/TEV-45779 High Dose | Transition Period: XOLAIR/TEV-45779 Low Dose
Number analyzed (Participants) | 170 | 91 | 91 | 46 | 93 | 47
units on a scale | -3.37 (6.641) [lower limit 6.641] | -2.66 (9.524) [lower limit 9.524] | -3.65 (7.953) [lower limit 7.953] | -2.54 (7.546) [lower limit 7.546] | -3.45 (8.387) [lower limit 8.387] | -3.12 (9.419) [lower limit 9.419]

16. Secondary Outcome: Change From Week 12 in the Physician's (In-clinic) Assessment of UAS7 at Week 24
Description: as for outcome 7
Time Frame: Week 12, Week 24
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Transition Period: TEV-45779/TEV-45779 High Dose | Transition Period: TEV-45779/TEV-45779 Low Dose | Transition Period: XOLAIR/XOLAIR High Dose | Transition Period: XOLAIR/XOLAIR Low Dose | Transition Period: XOLAIR/TEV-45779 High Dose | Transition Period: XOLAIR/TEV-45779 Low Dose
Number analyzed (Participants) | 175 | 91 | 93 | 49 | 92 | 48
units on a scale | -0.55 (1.556) [lower limit 1.556] | -0.40 (2.032) [lower limit 2.032] | -0.27 (1.360) [lower limit 1.360] | -0.53 (1.838) [lower limit 1.838] | -0.38 (1.413) [lower limit 1.413] | -0.67 (1.548) [lower limit 1.548]

17. Secondary Outcome: Change From Week 12 in the Weekly Number of Wheals Score at Weeks 24 and 40
Description: as for outcome 8
Time Frame: Week 12, Weeks 24 and 40
Population: The TITT analysis set included all participants re-randomized in the transition period. 'Overall number of participants analyzed' = participants evaluable for this endpoint. 'Number analyzed' = participants evaluable at specified timepoint.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Transition Period: TEV-45779/TEV-45779 High Dose | Transition Period: TEV-45779/TEV-45779 Low Dose | Transition Period: XOLAIR/XOLAIR High Dose | Transition Period: XOLAIR/XOLAIR Low Dose | Transition Period: XOLAIR/TEV-45779 High Dose | Transition Period: XOLAIR/TEV-45779 Low Dose
Number analyzed (Participants) | 170 | 91 | 91 | 46 | 93 | 47
units on a scale
  Change at Week 24 | -1.73 (3.649) | -1.29 (5.262) | -1.84 (4.139) | -1.33 (4.793) | -1.67 (4.510) | -1.03 (5.281)
  Change at Week 40: number analyzed (Participants) | 145 | 75 | 75 | 39 | 83 | 39
  Change at Week 40 | 1.87 (7.412) | 0.60 (8.236) | 1.53 (6.953) | 2.05 (6.110) | 2.77 (8.620) | 2.13 (7.809)

18. Secondary Outcome: Change From Week 12 in the Weekly Size of the Largest Wheals Score at Weeks 24 and 40
Description: The weekly size of the largest wheals score was calculated from eDiary data. A wheal score of 0 was assigned when <10 small wheals (diameter <3 cm) were present, presence of 10-50 small wheals or less than 10 large wheals (diameter >3 cm) was denoted by score 1. A score of 2 was assigned when more than 50 small wheals or 10 to 50 large wheals were present. A score of 3 denoted wheals covering almost the entire body surface area. A weekly score was defined as sum of available daily size of the largest wheals scores in that week, divided by the number of days for which a daily score was available, multiplied by 7. The possible range of the weekly score was therefore 0 (best score) to 21 (worst score) with higher scores indicating more severity.
Time Frame: Week 12, Weeks 24 and 40
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Transition Period: TEV-45779/TEV-45779 High Dose | Transition Period: TEV-45779/TEV-45779 Low Dose | Transition Period: XOLAIR/XOLAIR High Dose | Transition Period: XOLAIR/XOLAIR Low Dose | Transition Period: XOLAIR/TEV-45779 High Dose | Transition Period: XOLAIR/TEV-45779 Low Dose
Number analyzed (Participants) | 170 | 91 | 91 | 46 | 93 | 47
units on a scale
  Change at Week 24 | -1.87 (3.898) | -1.28 (4.697) | -1.78 (4.334) | -1.18 (4.464) | -1.94 (4.776) | -0.88 (4.456)
  Change at Week 40: number analyzed (Participants) | 145 | 75 | 75 | 39 | 83 | 39
  Change at Week 40 | 1.46 (7.434) | 0.72 (7.899) | 1.34 (7.332) | 2.35 (5.968) | 2.71 (8.706) | 1.87 (7.798)

19. Secondary Outcome: Percentage of Angioedema-Free Days From Week 12 to Week 24
Description: Percentage of angioedema-free days from Week 12 to Week 24 was calculated based on the diary data as the number of days in the diary between the dates of Week 12 and Week 24 visits with no angioedema episodes, divided by the total number of days with diary entries in this time span * 100%.
Time Frame: Week 12 to Week 24
Population: as for outcome 15
Measure: Median (Full Range); unit: percentage of days
Arm/Group | Transition Period: TEV-45779/TEV-45779 High Dose | Transition Period: TEV-45779/TEV-45779 Low Dose | Transition Period: XOLAIR/XOLAIR High Dose | Transition Period: XOLAIR/XOLAIR Low Dose | Transition Period: XOLAIR/TEV-45779 High Dose | Transition Period: XOLAIR/TEV-45779 Low Dose
Number analyzed (Participants) | 184 | 97 | 97 | 51 | 97 | 50
percentage of days | 100.00 (0.0) [0.0 to 100.0] | 100.00 (0.0) [0.0 to 100.0] | 100.00 (0.0) [0.0 to 100.0] | 100.00 (0.0) [0.0 to 100.0] | 100.00 (0.0) [0.0 to 100.0] | 100.00 (0.0) [0.0 to 100.0]

20. Secondary Outcome: Change From Week 12 in the Overall DLQI Score at Weeks 24 and 40
Description: as for outcome 13
Time Frame: Week 12, Weeks 24 and 40
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Transition Period: TEV-45779/TEV-45779 High Dose | Transition Period: TEV-45779/TEV-45779 Low Dose | Transition Period: XOLAIR/XOLAIR High Dose | Transition Period: XOLAIR/XOLAIR Low Dose | Transition Period: XOLAIR/TEV-45779 High Dose | Transition Period: XOLAIR/TEV-45779 Low Dose
Number analyzed (Participants) | 179 | 93 | 93 | 49 | 94 | 48
units on a scale
  Change at Week 24 | -1.44 (3.621) | -0.43 (5.619) | -1.19 (4.387) | -1.82 (5.552) | -0.88 (4.788) | -1.60 (4.271)
  Change at Week 40: number analyzed (Participants) | 160 | 83 | 85 | 41 | 86 | 42
  Change at Week 40 | 1.65 (7.581) | 1.05 (7.545) | 0.51 (7.096) | 0.39 (5.098) | 2.45 (7.791) | 1.10 (7.570)

21. Secondary Outcome: Number of Participants With at Least One Treatment-emergent Adverse Event (TEAE) in the Main Treatment Period
Description: An adverse event (AE) was defined as any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. Serious AEs (SAEs) were defined as death, a life-threatening AE, inpatient hospitalization or prolongation of existing hospitalization, persistent or significant disability or incapacity, a congenital anomaly or birth defect, or an important medical event that jeopardized participant and required medical intervention to prevent 1 of the outcomes listed in this definition. AEs were considered TEAEs if onset occurred or worsened on or after the first dose date. A summary of other non-serious AEs and all serious AEs, regardless of causality is located in Reported AE section.
Time Frame: Baseline up to Week 12
Population: The main treatment period safety analysis set included all randomized participants who received at least 1 dose of study drug during the main treatment period.
Measure: Count of Participants; unit: Participants
Arm/Group | Main Treatment Period: TEV-45779 High Dose | Main Treatment Period: TEV-45779 Low Dose | Main Treatment Period: XOLAIR High Dose | Main Treatment Period: XOLAIR Low Dose
Number analyzed (Participants) | 201 | 102 | 203 | 102
Participants | 64 | 37 | 71 | 33

22. Secondary Outcome: Number of Participants With at Least One TEAE Week 12 up to Week 24
Description: An AE was defined as any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. SAEs were defined as death, a life-threatening AE, inpatient hospitalization or prolongation of existing hospitalization, persistent or significant disability or incapacity, a congenital anomaly or birth defect, or an important medical event that jeopardized participant and required medical intervention to prevent 1 of the outcomes listed in this definition. AEs were considered TEAEs if onset occurred or worsened on or after the first dose date. A summary of other non-serious AEs and all serious AEs, regardless of causality is located in Reported AE section.
Time Frame: Week 12 up to Week 24
Population: The transition period safety analysis set included all randomized participants who received the study drug at Week 12.
Measure: Count of Participants; unit: Participants
Arm/Group | Transition Period: TEV-45779/TEV-45779 High Dose | Transition Period: TEV-45779/TEV-45779 Low Dose | Transition Period: XOLAIR/XOLAIR High Dose | Transition Period: XOLAIR/XOLAIR Low Dose | Transition Period: XOLAIR/TEV-45779 High Dose | Transition Period: XOLAIR/TEV-45779 Low Dose
Number analyzed (Participants) | 188 | 98 | 97 | 51 | 97 | 50
Participants | 78 | 34 | 43 | 18 | 38 | 16

23. Secondary Outcome: Number of Participants With Antidrug Antibodies (ADAs) in the Main Treatment Period
Description: Number of participants with positive ADA, positive ADA not treatment-related, and negative ADA are reported.
Time Frame: Baseline up to Week 12
Population: The main treatment period safety analysis set included all randomized participants who received at least 1 dose of study drug during the main treatment period. 'Overall number of participants analyzed' = participants with ADA status at any time during the main treatment period.
Measure: Count of Participants; unit: Participants
Arm/Group | Main Treatment Period: TEV-45779 High Dose | Main Treatment Period: TEV-45779 Low Dose | Main Treatment Period: XOLAIR High Dose | Main Treatment Period: XOLAIR Low Dose
Number analyzed (Participants) | 199 | 101 | 201 | 102
Participants
  Positive | 18 | 6 | 37 | 13
  Positive, Not Treatment Related | 8 | 5 | 5 | 4
  Negative | 173 | 90 | 159 | 85

24. Secondary Outcome: Number of Participants With ADAs From Week 12 to Week 24
Description: Number of participants with positive ADA, positive ADA not treatment-related, and negative ADA are reported.
Time Frame: Week 12 up to Week 24
Population: The transition period safety analysis set included all randomized participants who received the study drug at Week 12. 'Overall number of participants analyzed' = participants with ADA status at any time during the transition period.
Measure: Count of Participants; unit: Participants
Arm/Group | Transition Period: TEV-45779/TEV-45779 High Dose | Transition Period: TEV-45779/TEV-45779 Low Dose | Transition Period: XOLAIR/XOLAIR High Dose | Transition Period: XOLAIR/XOLAIR Low Dose | Transition Period: XOLAIR/TEV-45779 High Dose | Transition Period: XOLAIR/TEV-45779 Low Dose
Number analyzed (Participants) | 182 | 95 | 96 | 50 | 96 | 48
Participants
  Positive | 34 | 15 | 10 | 4 | 14 | 8
  Positive, Not Treatment Related | 6 | 4 | 3 | 1 | 1 | 2
  Negative | 142 | 76 | 83 | 45 | 81 | 38

ADVERSE EVENTS:
Time Frame: Baseline up to Week 40
Description: The safety analysis set included all randomized participants who received at least 1 dose of study drug. The transition period safety analysis set included all randomized participants who received the study drug at Week 12.
Groups:
- Main Treatment Period: TEV-45779 High Dose: Participants received TEV-45779 SC injection at a high dose level Q4W at Weeks 0, 4, and 8.
- Transition Period: TEV-45779/TEV-45779 High Dose: Participants who received TEV-45779 SC injection at a high dose level in the main treatment period continued to receive TEV-45779 at the same dose level at Weeks 12, 16, and 20 in the transition period.
- Transition Period: TEV-45779/TEV-45779 Low Dose: Participants who received TEV-45779 SC injection at a low dose level in the main treatment period continued to receive TEV-45779 at the same dose level at Weeks 12, 16, and 20 in the transition period.
- Transition Period: XOLAIR/XOLAIR High Dose: Participants who received XOLAIR SC injection at a high dose level in the main treatment period continued to receive XOLAIR at the same dose level at Weeks 12, 16, and 20 in the transition period.
- Transition Period: XOLAIR/XOLAIR Low Dose: Participants who received XOLAIR SC injection at a low dose level in the main treatment period continued to receive XOLAIR at the same dose level at Weeks 12, 16, and 20 in the transition period.
- Transition Period: XOLAIR/TEV-45779 High Dose: Participants who received XOLAIR SC injection at a high dose level in the main treatment period, received TEV-45779 at a high dose level at Weeks 12, 16, and 20 in the transition period.
- Transition Period: XOLAIR/TEV-45779 Low Dose: Participants who received XOLAIR SC injection at a low dose level in the main treatment period, received TEV-45779 at a low dose level at Weeks 12, 16, and 20 in the transition period.
Arm/Group | Main Treatment Period: TEV-45779 High Dose | Main Treatment Period: TEV-45779 Low Dose | Main Treatment Period: XOLAIR High Dose | Main Treatment Period: XOLAIR Low Dose | Transition Period: TEV-45779/TEV-45779 High Dose | Transition Period: TEV-45779/TEV-45779 Low Dose | Transition Period: XOLAIR/XOLAIR High Dose | Transition Period: XOLAIR/XOLAIR Low Dose | Transition Period: XOLAIR/TEV-45779 High Dose | Transition Period: XOLAIR/TEV-45779 Low Dose
All-Cause Mortality (participants affected / at risk) | 0/201 | 0/102 | 0/203 | 0/102 | 0/188 | 0/98 | 0/97 | 0/51 | 0/97 | 0/50
Serious Adverse Events (participants affected / at risk) | 1/201 | 0/102 | 3/203 | 0/102 | 4/188 | 3/98 | 4/97 | 0/51 | 1/97 | 1/50
Other Adverse Events (participants affected / at risk) | 30/201 | 19/102 | 30/203 | 10/102 | 29/188 | 11/98 | 16/97 | 8/51 | 10/97 | 6/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Main Treatment Period: TEV-45779 High Dose (N=201) | Main Treatment Period: TEV-45779 Low Dose (N=102) | Main Treatment Period: XOLAIR High Dose (N=203) | Main Treatment Period: XOLAIR Low Dose (N=102) | Transition Period: TEV-45779/TEV-45779 High Dose (N=188) | Transition Period: TEV-45779/TEV-45779 Low Dose (N=98) | Transition Period: XOLAIR/XOLAIR High Dose (N=97) | Transition Period: XOLAIR/XOLAIR Low Dose (N=51) | Transition Period: XOLAIR/TEV-45779 High Dose (N=97) | Transition Period: XOLAIR/TEV-45779 Low Dose (N=50)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Strangulated umbilical hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epiglottitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Erysipelas (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyelonephritis chronic (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lower limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chondromalacia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Adenomyosis (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Main Treatment Period: TEV-45779 High Dose (N=201) | Main Treatment Period: TEV-45779 Low Dose (N=102) | Main Treatment Period: XOLAIR High Dose (N=203) | Main Treatment Period: XOLAIR Low Dose (N=102) | Transition Period: TEV-45779/TEV-45779 High Dose (N=188) | Transition Period: TEV-45779/TEV-45779 Low Dose (N=98) | Transition Period: XOLAIR/XOLAIR High Dose (N=97) | Transition Period: XOLAIR/XOLAIR Low Dose (N=51) | Transition Period: XOLAIR/TEV-45779 High Dose (N=97) | Transition Period: XOLAIR/TEV-45779 Low Dose (N=50)
Injection site erythema (General disorders) | 15 (24) | 10 (14) | 13 (21) | 7 (12) | 8 (17) | 5 (6) | 3 (4) | 2 (3) | 6 (9) | 3 (8)
Injection site induration (General disorders) | 12 (17) | 6 (6) | 12 (15) | 5 (7) | 7 (15) | 3 (4) | 3 (4) | 1 (1) | 3 (5) | 3 (9)
Injection site pain (General disorders) | 13 (30) | 9 (11) | 11 (21) | 5 (11) | 8 (14) | 3 (7) | 2 (2) | 2 (4) | 1 (2) | 2 (6)
Injection site swelling (General disorders) | 9 (10) | 4 (4) | 4 (4) | 3 (4) | 6 (9) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 3 (8)
COVID-19 (Infections and infestations) | 5 (5) | 5 (5) | 8 (8) | 0 (0) | 9 (9) | 5 (5) | 7 (7) | 3 (3) | 1 (1) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 5 (5) | 3 (4) | 2 (2) | 0 (0) | 9 (11) | 1 (1) | 5 (5) | 2 (2) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor has the right 60 days before submission for publication to review/provide comments. If the Sponsor's review shows that potentially patentable subject matter would be disclosed, publication or public disclosure shall be delayed for up to 90 additional days in order for the Sponsor, or Sponsor's designees, to file the necessary patent applications. In multicenter trials, each PI will postpone single center publications until after disclosure or publication of multicenter data.

DOCUMENTS (2):
  • Study Protocol (2023-02-15): https://cdn.clinicaltrials.gov/large-docs/92/NCT04976192/Prot_000.pdf
  • Statistical Analysis Plan (2024-01-02): https://cdn.clinicaltrials.gov/large-docs/92/NCT04976192/SAP_001.pdf